CLINICAL TRIAL: NCT02418312
Title: Efficacy of H2 Receptor Antagonist in Prevention of Thienopyridine-related Peptic Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Ping-I (William) Hsu, M.D., Professor, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VGHKS11-CT12-10
Record Dates: First submitted 2015-04-12; First posted 2015-04-16 (Estimated); Results first posted 2019-03-11 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Peptic Ulcer
Keywords: histamine-2 receptor antagonist; peptic ulcer; thienopyridine; prevention
MeSH Terms: conditions — Peptic Ulcer | interventions — Histamine H2 Antagonists; Famotidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- histamine-2 receptor antagonist group (Active Comparator): famotidine 40mg qd for 6 months.
  Interventions: Drug: histamine-2 receptor antagonist
- placebo group (Placebo Comparator): placebo for 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: histamine-2 receptor antagonist — famotidine 40 mg qd plus thienopyridine
  Other Names: famotidine 40 mg qd
  Arms: histamine-2 receptor antagonist group
Drug: Placebo — placebo plus thienopyridine
  Arms: placebo group

SUMMARY:
Whether H2 receptor antagonist can prevent thienopyridine-related peptic ulcer remains unclear.

DETAILED DESCRIPTION:
The aim of the prospective, randomized study is investigate the efficacy of H2 receptor antagonist in prevention of thienopyridine-related peptic ulcer and gastrointestinal bleeding in patients with an ulcer history. We plan to enroll 236 thienopyridine (clopidogrel or ticlopidine) users with a peptic ulcer history who don't have baseline gastroduodenal ulcers at initial endoscopy . The patients will be randomly assigned to receive either (1) famotidine (40 mg qd) plus thienopyridine used previously or (2) placebo plus thienopyridine treatment alone for 6 months. The ulcer recurrence rate between the treatment gruops will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. The past history of gastroduodenal ulcer and underwent endoscopy for dyspeptic symptoms.
2. thienopyridine users without baseline gastroduodenal ulcer at initial endoscopy.
3. They are adult patients aged least 20 years of age.

Exclusion Criteria:

1. They have a history of gastric or duodenal surgery other than oversewing of a perforation.
2. They require long-term treatment with non-steroidal anti-inflammatory drugs.
3. serious disease.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2012-01; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ping-I Hsu, Bachelor, Study Chair — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Savi P, Nurden P, Nurden AT, Levy-Toledano S, Herbert JM. Clopidogrel: a review of its mechanism of action. Platelets. 1998;9(3-4):251-5. doi: 10.1080/09537109876799. PMID 16793712
- [Background] Boeynaems JM, van Giezen H, Savi P, Herbert JM. P2Y receptor antagonists in thrombosis. Curr Opin Investig Drugs. 2005 Mar;6(3):275-82. PMID 15816504
- [Background] Yusuf S, Zhao F, Mehta SR, Chrolavicius S, Tognoni G, Fox KK; Clopidogrel in Unstable Angina to Prevent Recurrent Events Trial Investigators. Effects of clopidogrel in addition to aspirin in patients with acute coronary syndromes without ST-segment elevation. N Engl J Med. 2001 Aug 16;345(7):494-502. doi: 10.1056/NEJMoa010746. PMID 11519503
- [Background] Bhatt DL, Fox KA, Hacke W, Berger PB, Black HR, Boden WE, Cacoub P, Cohen EA, Creager MA, Easton JD, Flather MD, Haffner SM, Hamm CW, Hankey GJ, Johnston SC, Mak KH, Mas JL, Montalescot G, Pearson TA, Steg PG, Steinhubl SR, Weber MA, Brennan DM, Fabry-Ribaudo L, Booth J, Topol EJ; CHARISMA Investigators. Clopidogrel and aspirin versus aspirin alone for the prevention of atherothrombotic events. N Engl J Med. 2006 Apr 20;354(16):1706-17. doi: 10.1056/NEJMoa060989. Epub 2006 Mar 12. PMID 16531616
- [Background] Mehta SR, Yusuf S, Peters RJ, Bertrand ME, Lewis BS, Natarajan MK, Malmberg K, Rupprecht H, Zhao F, Chrolavicius S, Copland I, Fox KA; Clopidogrel in Unstable angina to prevent Recurrent Events trial (CURE) Investigators. Effects of pretreatment with clopidogrel and aspirin followed by long-term therapy in patients undergoing percutaneous coronary intervention: the PCI-CURE study. Lancet. 2001 Aug 18;358(9281):527-33. doi: 10.1016/s0140-6736(01)05701-4. PMID 11520521
- [Background] CAPRIE Steering Committee. A randomised, blinded, trial of clopidogrel versus aspirin in patients at risk of ischaemic events (CAPRIE). CAPRIE Steering Committee. Lancet. 1996 Nov 16;348(9038):1329-39. doi: 10.1016/s0140-6736(96)09457-3. PMID 8918275
- [Background] Fork FT, Lafolie P, Toth E, Lindgarde F. Gastroduodenal tolerance of 75 mg clopidogrel versus 325 mg aspirin in healthy volunteers. A gastroscopic study. Scand J Gastroenterol. 2000 May;35(5):464-9. doi: 10.1080/003655200750023705. PMID 10868447
- [Background] Ng FH, Wong SY, Chang CM, Chen WH, Kng C, Lanas AI, Wong BC. High incidence of clopidogrel-associated gastrointestinal bleeding in patients with previous peptic ulcer disease. Aliment Pharmacol Ther. 2003 Aug 15;18(4):443-9. doi: 10.1046/j.1365-2036.2003.01693.x. PMID 12940930
- [Background] Chan FK, Ching JY, Hung LC, Wong VW, Leung VK, Kung NN, Hui AJ, Wu JC, Leung WK, Lee VW, Lee KK, Lee YT, Lau JY, To KF, Chan HL, Chung SC, Sung JJ. Clopidogrel versus aspirin and esomeprazole to prevent recurrent ulcer bleeding. N Engl J Med. 2005 Jan 20;352(3):238-44. doi: 10.1056/NEJMoa042087. PMID 15659723
- [Background] Ma L, Elliott SN, Cirino G, Buret A, Ignarro LJ, Wallace JL. Platelets modulate gastric ulcer healing: role of endostatin and vascular endothelial growth factor release. Proc Natl Acad Sci U S A. 2001 May 22;98(11):6470-5. doi: 10.1073/pnas.111150798. Epub 2001 May 15. PMID 11353854
- [Background] Hsu PI, Lai KH, Liu CP. Esomeprazole with clopidogrel reduces peptic ulcer recurrence, compared with clopidogrel alone, in patients with atherosclerosis. Gastroenterology. 2011 Mar;140(3):791-8. doi: 10.1053/j.gastro.2010.11.056. Epub 2010 Dec 7. PMID 21144850
- [Background] Laine L, Hennekens C. Proton pump inhibitor and clopidogrel interaction: fact or fiction? Am J Gastroenterol. 2010 Jan;105(1):34-41. doi: 10.1038/ajg.2009.638. Epub 2009 Nov 10. PMID 19904241
- [Background] Sibbing D, Kastrati A. Risk of combining PPIs with thienopyridines: fact or fiction? Lancet. 2009 Sep 19;374(9694):952-954. doi: 10.1016/S0140-6736(09)61562-2. Epub 2009 Aug 31. No abstract available. PMID 19726077
- [Background] Gilard M, Arnaud B, Cornily JC, Le Gal G, Lacut K, Le Calvez G, Mansourati J, Mottier D, Abgrall JF, Boschat J. Influence of omeprazole on the antiplatelet action of clopidogrel associated with aspirin: the randomized, double-blind OCLA (Omeprazole CLopidogrel Aspirin) study. J Am Coll Cardiol. 2008 Jan 22;51(3):256-60. doi: 10.1016/j.jacc.2007.06.064. PMID 18206732
- [Background] Simon T, Verstuyft C, Mary-Krause M, Quteineh L, Drouet E, Meneveau N, Steg PG, Ferrieres J, Danchin N, Becquemont L; French Registry of Acute ST-Elevation and Non-ST-Elevation Myocardial Infarction (FAST-MI) Investigators. Genetic determinants of response to clopidogrel and cardiovascular events. N Engl J Med. 2009 Jan 22;360(4):363-75. doi: 10.1056/NEJMoa0808227. Epub 2008 Dec 22. PMID 19106083
- [Background] Ho PM, Maddox TM, Wang L, Fihn SD, Jesse RL, Peterson ED, Rumsfeld JS. Risk of adverse outcomes associated with concomitant use of clopidogrel and proton pump inhibitors following acute coronary syndrome. JAMA. 2009 Mar 4;301(9):937-44. doi: 10.1001/jama.2009.261. PMID 19258584
- [Background] Juurlink DN, Gomes T, Ko DT, Szmitko PE, Austin PC, Tu JV, Henry DA, Kopp A, Mamdani MM. A population-based study of the drug interaction between proton pump inhibitors and clopidogrel. CMAJ. 2009 Mar 31;180(7):713-8. doi: 10.1503/cmaj.082001. Epub 2009 Jan 28. PMID 19176635
- [Background] Taha AS, Hudson N, Hawkey CJ, Swannell AJ, Trye PN, Cottrell J, Mann SG, Simon TJ, Sturrock RD, Russell RI. Famotidine for the prevention of gastric and duodenal ulcers caused by nonsteroidal antiinflammatory drugs. N Engl J Med. 1996 May 30;334(22):1435-9. doi: 10.1056/NEJM199605303342204. PMID 8618582
- [Background] Hudson N, Taha AS, Russell RI, Trye P, Cottrell J, Mann SG, Swanell AJ, Sturrock RD, Hawkey CJ. Famotidine for healing and maintenance in nonsteroidal anti-inflammatory drug-associated gastroduodenal ulceration. Gastroenterology. 1997 Jun;112(6):1817-22. doi: 10.1053/gast.1997.v112.pm9178671.
- [Background] Taha AS, Dahill S, Morran C, Hudson N, Hawkey CJ, Lee FD, Sturrock RD, Russell RI. Neutrophils, Helicobacter pylori, and nonsteroidal anti-inflammatory drug ulcers. Gastroenterology. 1999 Feb;116(2):254-8. doi: 10.1016/s0016-5085(99)70120-4. PMID 9922304
- [Background] Taha AS, McCloskey C, Prasad R, Bezlyak V. Famotidine for the prevention of peptic ulcers and oesophagitis in patients taking low-dose aspirin (FAMOUS): a phase III, randomised, double-blind, placebo-controlled trial. Lancet. 2009 Jul 11;374(9684):119-25. doi: 10.1016/S0140-6736(09)61246-0. Epub 2009 Jul 3. PMID 19577798
- [Background] Ng FH, Wong SY, Lam KF, Chu WM, Chan P, Ling YH, Kng C, Yuen WC, Lau YK, Kwan A, Wong BC. Famotidine is inferior to pantoprazole in preventing recurrence of aspirin-related peptic ulcers or erosions. Gastroenterology. 2010 Jan;138(1):82-8. doi: 10.1053/j.gastro.2009.09.063. Epub 2009 Nov 11. PMID 19837071
- [Background] Hsu PI, Lai KH, Wu CJ, Tseng HH, Tsay FW, Peng NJ, Chen TA, Chuah SK, Lin WS, Lo GH. High-dose versus low-dose esomeprazole-based triple therapy for Helicobacter pylori infection. Eur J Clin Invest. 2007 Sep;37(9):724-30. doi: 10.1111/j.1365-2362.2007.01852.x. PMID 17696962

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Histamine-2 Receptor Antagonist Group | Placebo Group
Started | 114 | 114
Completed | 114 | 114
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Histamine-2 Receptor Antagonist Group | Placebo Group | Total
Number analyzed (Participants) | 114 | 114 | 228
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.7 (11.9) | 72.9 (11.1) | 72.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 36 | 64
  Male | 86 | 78 | 164
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 114 | 114 | 228
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
history of smoking [Number; unit: participants] | 14 | 10 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Healed Peptic Ulcer
Description: Follow-up endoscopy was performed at the end of the 6th month
Time Frame: 6 months
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | Histamine-2 Receptor Antagonist Group | Placebo Group
Number analyzed (Participants) | 114 | 114
participants | 106 | 101

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Histamine-2 Receptor Antagonist Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/114 | 0/114
Serious Adverse Events (participants affected / at risk) | 0/114 | 0/114
Other Adverse Events (participants affected / at risk) | 3/114 | 2/114
OTHER ADVERSE EVENTS (reported when occurring in more than 1.3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Histamine-2 Receptor Antagonist Group (N=114) | Placebo Group (N=114)
skin rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
persistent dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The trial was performed in a single country

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-09): https://cdn.clinicaltrials.gov/large-docs/12/NCT02418312/Prot_SAP_000.pdf